CLINICAL TRIAL: NCT06152003
Title: Developing and Piloting a Multilevel Intervention to Address Psychosocial and Structural Syndemics in People With HIV in South Africa
Brief Title: Intervention Development for Syndemics Among PWH in SA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Cape Town (Other); University of Miami (Other); University of the Western Cape (Other); University of Stellenbosch (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P002344
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: Syndemic Problems; ART Adherence; Food Insecurity; Depression; Post-traumatic Stress Disorder
MeSH Terms: conditions — HIV Infections; Depression; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Syndemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent assessors will be used to measure study outcomes of the RCT at follow-up assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment as Usual (ETAU) (No Intervention): We anticipate the control condition will contain the following: the enhanced treatment as usual (ETAU; n=30) will consist of PWH receiving treatment at their HIV primary care clinic as usual, enhanced by supplemental food parcels and referrals for mental health care and food service organizations. Treatment as usual for mental health care is evaluation by a nurse and referral to a medical officer or to a traveling psychologist available 1 day per week. Because there is no standard of care for food insecurity, we propose that all participants will receive food parcels, but ETAU participants will not receive case management or psychosocial intervention.
- Cognitive Behavioral Therapy for Syndemics and Adherence (CBT-SA) (Experimental): We anticipate the intervention condition (CBT-SA) will contain the following: cognitive behavioral therapy for syndemics and adherence (CBT-SA; n=30) likely will be comprised of both psychosocial and structural intervention components, based on the results of Aim 1 and refinement in Aim 2. In addition to food parcels, we expect the CBT-SA condition will also receive nutritional counseling, linkage to care, and case management. Only the CBT-SA condition will receive the psychological intervention for depression and PTSD and adherence counseling. Specific intervention components will be informed by prior aims.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Syndemics and Adherence (CBT-SA)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Syndemics and Adherence (CBT-SA) — We anticipate the intervention will contain the following: CBT for depression and trauma, Life-Steps for ART adherence, nutritional counseling, supplementary food parcels, case management, linkage to care. Specific intervention components will be informed by prior aims.
  Arms: Cognitive Behavioral Therapy for Syndemics and Adherence (CBT-SA)

SUMMARY:
In South Africa, the country with the highest HIV prevalence (19%), co-occurring problems such as depression, post-traumatic stress, and food insecurity interact to enhance one another (i.e., syndemic problems) and are associated with worse HIV outcomes such as worse antiretroviral therapy (ART) adherence and worse viral load. This study proposes to: 1) explore how syndemic problems work together to make health worse for people with HIV (PWH) and explore what people think about a potential treatment; 2) develop a treatment to address syndemic problems and improve ART adherence (CBT-SA); 3a) assess whether people are willing to receive the CBT-SA we it can actually be done; and 3b) identify factors that make it easier or more difficult to receive CBT-SA.

DETAILED DESCRIPTION:
South Africa (SA) has a generalized HIV epidemic, and the highest HIV prevalence rate (19%). Psychosocial (e.g., depression, post-traumatic stress) and structural problems (e.g., food insecurity) are associated with worse antiretroviral therapy (ART) adherence and higher viral load. Depression, post-traumatic stress, and food insecurity are also highly comorbid and are thought to interact synergistically to confer greater risk for worse HIV outcomes (i.e., syndemic problems). The proposed specific aims are to: 1) explore the complex interrelationships between food insecurity, depression, and post-traumatic stress, as they relate to engagement in HIV care, and explore attitudes to potential intervention components; 2) develop a multilevel intervention to address syndemic problems and improve adherence (CBT-SA) and conduct an iterative proof-of-concept pilot trial use syndemic theory; 3a) assess the feasibility and acceptability of CBT-SA in a pilot RCT; and 3b) identify barriers and facilitators of CBT-SA engagement among PWH and uptake among care providers and other key local partners to inform a future hybrid effectiveness/implementation R01 trial. If successful, this intervention would be further tested for effectiveness and implementation in a future application.

ELIGIBILITY:
Inclusion Criteria:

1. Patient receiving HIV care in Khayelitsha (confirmed by medical record)
2. Currently prescribed TDF-based ART, with recent difficulties with ART adherence (self-reported in past 30 days / confirmed by pharmacy refill data)
3. Mild, moderate, or severe food insecurity (measured by HFIAS categories) AND ≥1 of the following:

   * Clinically significant depressive symptoms (CES-D ≥ 16)
   * Clinically significant post-traumatic stress symptoms (SPAN ≥ 5)
4. 18 years of age or older

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. In the past year: received CBT for depression or PTSD, or received supplemental food parcels or nutritional counseling
3. Current untreated or undertreated serious mental health issue that would interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
75% of participants randomized to CBT-SA attend at least 66% of the sessions | 6-month follow-up
  We will calculate the percentage of participants randomized to the CBT-SA condition who attend 66% or greater of the total number of sessions. CBT-SA will be considered feasible and acceptable if 75% of the participants attend 66% or more of the sessions.
75% of the participants randomized to CBT-SA attend the 6-month follow-up visit. | 6-month follow-up
  We will calculate the percentage of participants randomized to the CBT-SA condition who attend the 6-month follow-up visit. CBT-SA will be considered feasible and acceptable if 75% of the participants attend the 6-month follow-up visit.

SECONDARY OUTCOMES:
ART adherence | 6-month follow-up
  ART adherence via dried blood spots on TDF-based regimens
Presence of depression measured by the DIAMOND diagnostic instrument | 6-month follow-up
  Whether participants meet criteria or not on the depression module of the DIAMOND Diagnostic Measure.
Presence of PTSD measured by the DIAMOND diagnostic instrument | 6-month follow-up
  Whether participants meet criteria or not on the PTSD module of the DIAMOND Diagnostic Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Conall O'Cleirigh, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
In accordance with our DMS plan, public use study data will be deposited to the Inter-university Consortium for Political and Social Research (ICPSR). ICPSR is a CoreTrustSeal certified repository providing long-term access to and preservation of data packages curated by domain specialists.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available one year after we have achieved the main aims of the project (i.e., publication of the main outcome papers). ICPSR will make decisions about how long to preserve the data; however, ICPSR permanently archives deposited files.
Access Criteria: TBD.